CLINICAL TRIAL: NCT06507462
Title: Construction and Validation of a Diagnostic Prediction Model for Prostate Cancer in Patients With PI-RADS Score 3: a Multicenter, Retrospective Study
Brief Title: A Diagnostic Prediction Model for Prostate Cancer in Patients With PI-RADS Score 3
Status: Completed | Type: Observational
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, XiaoJun, Professor, Anhui Provincial Hospital
Other Study IDs: 2024-ky312
Record Dates: First submitted 2024-07-04; First posted 2024-07-18 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Predictive model; Diagnosis; Prostate Imaging-Reporting and Data System
MeSH Terms: conditions — Prostatic Neoplasms; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with clinical suspicion of prostate cancer and have PI-RADS score of 3: Patients with clinical suspicion of prostate cancer (see inclusion criteria) and have PI-RADS score (results of mpMRI) of 3.
  Interventions: Procedure: prostate biopsy

INTERVENTIONS:
Procedure: prostate biopsy — All patients were required to underwent transperineal prostate biopsy and have corresponding pathological diagnosis results.

SUMMARY:
The goal of this observational study is to construct a predictive model for improving the diagnostic accuracy in patients with PI-RADS score of 3. The main aims of this study are:

* Construct a diagnostic model of patients with PI-RADS of score.
* Internal and external validation of the model.
* Decision curve analysis. The data of participants was collected retrospectively.

DETAILED DESCRIPTION:
For patients with a PI-RADS score of 3, the diagnosis of prostate cancer is still use prostate biopsy, but the detection rates of prostate cancer and clinically significant prostate cancer are approximately 30% and 15%. It can be seen that most patients with PI-RADS 3 undergo unnecessary prostate biopsy and bear the risk of complications such as urinary tract infection. This makes most patients with PI-RADS 3 choose to refuse invasive prostate biopsy. Although researchers are committed to exploring biomarkers with high sensitivity and specificity, the application of biomarkers alone often cannot achieve the expected results. At present, the guidelines have recommended the use of diagnostic prediction models to assess patients' prostate cancer risk. Doctors and patients use diagnostic models to assess the risk of prostate cancer before prostate biopsy. For patients with a low probability of cancer, biopsy can be temporarily avoided, which to a certain extent reduces the phenomenon of prostate cancer overdiagnosis. This study plans to work with multiple medical centers to conduct statistical analysis based on existing prostate cancer screening markers combined with patients' clinical data such as prostate volume, prostate-specific antigen density, apparent diffusion coefficient, PI-RADS score and postoperative Gleason score, and then construct a prostate cancer diagnostic model to improve the diagnostic accuracy of prostate cancer for patients with PI-RADS score of 3. This will be of great significance for improving the early diagnosis of patients with PI-RADS 3 and reducing unnecessary prostate puncture biopsies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinically suspected prostate cancer (abnormal PSA level or DRE);
2. All patients have undergone mpMRI and have complete imaging data;
3. The PI-RADS score of patients was 3;
4. Prostate biopsy was performed and has clear pathological results.

Exclusion Criteria:

1. The patient's serum tPSA is <4ng/ml or >100ng/ml;
2. Repeated prostate biopsy;
3. The patient's clinical, imaging, or pathological data are incomplete.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a multicenter retrospective study. All enrolled patients were clinically suspected of prostate cancer (abnormal serum PSA level or DRE), had an indication for prostate biopsy and eventually underwent prostate biopsy. Before biospy, patients also need to complete mpMRI examination, the examination sequence includes at least multi-plane T2WI and multi-b value DWI, and the final patient PI-RADS score needs to be 3.
Sampling Method: Non-Probability Sample
Enrollment: 460 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Multivariate logistic regression analyses and calculate the odds ratios (95% confidence interval ) of the clinical variables for clinically significant prostate cancer | through study completion, an average of 3 months
  The clinically significant prostate cancer was defined as Gleason score ≥ 3+4

SECONDARY OUTCOMES:
Validation by calculating the C-statistics, drawing ROC curves (AUC values) and calibration curves. | through study completion, an average of 3 months
  Evaluate the discrimination and calibration of the model constructed by logistic regression analyses

CONTACTS AND LOCATIONS:
Overall Officials: Jun Xiao, Pro., Principal Investigator — The First Affiliated Hospital of USTC
Locations (3):
- China (3):
  - Department of Urology, The First Affiliated Hospital of Bengbu Medical University, Bengbu, Anhui
  - Department of Urology, The First Affiliated Hospital of USTC, Hefei, Anhui
  - Department of Urology, The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui

IPD SHARING:
Plan to Share IPD: Undecided